CLINICAL TRIAL: NCT06432517
Title: Identification of the Sources and Mechanisms of Energy Compensation in Humans
Brief Title: Sources and Mechanisms of Energy Compensation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Chief scientist, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SIAT-IRB-230515-H0653
Record Dates: First submitted 2024-04-02; First posted 2024-05-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Energy Expenditure; Exercise; Energy Intake; Food Preferences
Keywords: Energy compensation; Energy balance; Food Preferences
MeSH Terms: conditions — Motor Activity; Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Moderate to high intensity exercise (Experimental): BMI≥18.5, age between 18-40 years old, 81subjects.
  Interventions: Other: Power Bike（Ergoselect 100P）

INTERVENTIONS:
Other: Power Bike（Ergoselect 100P） — Changes in the participants' energy balance will be measured through moderate to high intensity exercise. Observation of food intake, body composition, metabolic rate, food assimilation rate.

SUMMARY:
Excess energy, obesity and obesity-related diseases are important global health issues. Although it is known that obesity is an issue of energy balance, the components of energy expenditure seem to be inter-related in complex non-additive ways. The aim of this study is to explore the downstream impacts of exercise on short term changes in both expenditure and energy intake. The primary question the investigators are asking is whether moderate to high intensity exercise influences the basal energy expenditure and/or energy intake/macronutrient preference in young adult males? (A similar study will be performed on females in a different registration). The investigators will use a specially designed feeding table to measure energy intake and macronutrient intake, which is easy to quantify intake compensation. Basal metabolism will be measured by hood indirect calorimetry. The investigators will explore the factors that influence the level of compensation in expenditure and intake, in particular body composition. Participants will be asked to come to the lab after 10 hours fast for body composition tests including Dual Energy X-ray Absorptiometry(DXA), Magnetic Resonance Image(MRI) and Bioelectrical Impedance Analysis(BIA). They will then be asked (not) to do 30 minutes of moderate-to-vigorous exercise after an energy-limiting breakfast, during which metabolic rate levels and changes in dietary composition will be recorded by gas exchange and standardized buffet. In addition, participants' subjective hunger and preferences will also be recorded by questionnaires. Venous blood will be collected to measure metabolic and hormone factors, blood glucose will be measured by Continuous Blood Glucose Monitor (CGM).

DETAILED DESCRIPTION:
81 participants will be recruited by posters and Wechat. The sample size is calculated using the paired t-test in power analysis, in which α value is 0.05, β value is 0.8, standard deviation is 372 (calculated from the energy intake data in the preliminary trial), and the difference is 108. The alternative hypothesis is greater than 108. The experiment lasted for 14 days, of which two and a half days will be carried out in the laboratory, and the other time only need to wear devices and live freely, which will not affect the normal life. The experiment is mainly divided into three parts:

1. Body composition: Items include weight, height, body fat mass (MRI), bone mass (DAX), body density (BODPOD), lean mass (MRI) and 3D parameters (3D scan). The participants will be required to fasting for at least 10 hours. After the test, they will be equipped with continuous glucose monitoring equipment (CGM), motion monitoring equipment (GT3X) and ambient temperature monitoring equipment (ibutton).
2. Controlled trial: The specific detection contents include resting energy expenditure (REE), active energy expenditure (AEE) and energy intake. The investigators will provide participants with three meals, as an energy restricted breakfast, a standard lunch and supper for dietary component testing. The subjective hunger and eating preference rate of participants will be measured by Visual Analogue Scale (VAS) and questionnaires. Non-physical activities such as working, reading and watching movies will be allowed during the experiment. Venous blood will be collected at several specific points (fasting 10 hours, after breakfast, before lunch and after lunch). In addition, sweat, urine and feces will also be collected.
3. Exercise trial: The schedule is the same as the control trial except for Blood drawing time and 30 minutes of power bike after breakfast, the intensity is 100 watt with 1 minute 25 watt break every 5 minute during the exercise. Venous blood will be collected at several specific points in time (just after exercise, before lunch and after lunch).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (men)
* 18-40 years old
* BMI (body mass index)≥18.5 kg/m2

Exclusion Criteria:

* Those who have undergone surgery in the past 6 months.
* People are requiring long-term medication.
* People have metabolic diseases, like diabetes, hypoglycemia, gout, osteoporosis, et al.
* People have digestive diseases, like gastric ulcer, pancreatitis, Intestinal obstruction, et al.
* People have sports injury, like fracture, Joint injury, et al.
* Those who have recently lost weight for various medical reasons (e.g. cancer, etc.).
* People are losing weight by tablets.
* People are suffering from infectious diseases (e.g. HIV, etc.)
* People have blood phobia, pathological hypo or hyper tension.
* People with impaired glucose tolerance.
* Those who are afflicted with claustrophobia.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Macronutrient preference | During lunchtime and dinnertime on both the control day(baseline) and exercise day(the day after control day), each test lasting for 40 minutes.
  Macronutrients preference will be recorded by the feeding table, macronutrient preference will be calculated in percentage(%).
Energy intake | During lunchtime and dinnertime on both the control day(baseline) and exercise day(the day after control day), each test lasting for 40 minutes.
  Response on standard feeding table, the food consumption will be recorded continuously by balances underneath each food dish. The total energy intake will be calculated in kilojoule (KJ).
Basal metabolic rate | The detection time spans over two days, the control day and the exercise day, from 8:00 am to 5:00 pm, with tests being conducted every hour and each test lasting for half an hour.
  Resting energy expenditure will be measured using indirect calorimetry via a respiratory hood system (Cosmed). The subject attends in the lab after an overnight fast. The person lies down on a flat bed and the hood is placed over their head. Metabolic rate (oxygen consumption and carbon dioxide production) are monitored for 40 minutes. The last 10 minutes is used as the measurement. Calorimeters will be assessed with a turbine test to ensure accuracy of measurements. Validation via an alcohol burn will be performed monthly.

SECONDARY OUTCOMES:
Blood glucose | Wear it for a total of 4 consecutive days, including the physical examination day, the control day, the exercise day, and the day following the exercise day.
  Blood glucose will be recorded by the continuous glucose monitoring system(CGM) in mmol/L.
Physical activity | Wear it for 14 days from the physical examination day
  Physical activity of the participants will be recorded using GT3X accelerometer worn near the hip for a consecutive period of 14 days. The monitor should not be worn while bathing or swimming. The first day is discarded along with any day where the wear time is less than 12 hours. For a valid measure the goal is to get 2 weekday and 2 weekend days.
Ambient temperature | Wear it for 14 days from the physical examination day
  The iButton (DS1921G) monitors will be provided for the assessment of both indoor and outdoor temperature of their living environment in centigrade(℃). The iButtons can be affixed to the hand bag (or clothes) to measure the subject exposure temperature, an indoor wall of home and workplace, and the building outside to measure the outdoor temperature using a strip of adhesive, water resistant, medical grade tape.
Circulating Biochemical indexes and hormones | The venous blood of volunteers will be collected 10 times on control and exercise days. (Control day: fasting, 1,2,3,4 hours after breakfast and 2 hours after lunch. Exercise day: 0,1,2 hours after exercise and 2 hours after lunch)
  Levels of circulating hormones (including leptin, insulin, ghrelin etc) will be measured when fasted and after a standard intervention meal. Levels of circulating hormones in the serum will be measured by ELISA (Bio Tek, Synergy4) in mmol/L.
Exercise | 30 minutes after breakfast(only on the exercise day), it last for 39 minutes, 30 minutes at 100 watts and 9 minutes at 25 watts.
  Physical activity will be carried out by the Ergoselect 100P(Power bike) at 100 watts
Exercise metabolic rate | 30 minutes after breakfast(only on the exercise day), it last for 39 minutes, 30 minutes at 100 watts and 9 minutes at 25 watts.
  Basal metabolic rate will be recorded by the Quark PFT ergo, The energy expenditure will be calculated in kilojoule (kj).
Weight | On the first morning of the experiment, it last for 10 minutes.
  Volunteers will be asked to fast for 10 hours and measured fasting weight (kilogram, kg) with light clothes and no shoes.
Height | On the first morning of the experiment, it last for 10 minutes.
  Height will be measured by seca 217 stable stadiometer in meter(m).
Waist circumferences | On the first morning of the experiment, it last for 15 minutes.
  Waist circumferences will be measured using a whole body laser scanner in centimeter(cm).
Hip circumferences | On the first morning of the experiment, it last for 15 minutes.
  Hip circumferences will be measured using a whole body laser scanner in centimeter(cm).
Bone mineral density | On the first morning of the experiment, it last for 8 minutes.
  Bone mineral density will be measured by Dual Energy X-ray Absorptiometry (Horizon Wi).
Fat mass | On the first morning of the experiment, it last for 30 minutes.
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ). and Bioimpedance Analysis (Tanita, MC-980).
Fat free mass | On the first morning of the experiment, it last for 30 minutes.
  Fat free mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ). and Bioimpedance Analysis (Tanita, MC-980).
Blood pressure | On both the control and exercise days, blood pressure will be measured prior to the basic energy expenditure(≈8:00 am), it last for 5 minutes.
  Systolic and diastolic blood pressure will be measured using an Omron sphygmomanometer.
Body temperature | On both the control and exercise days, the change of body temperature will be measured during lunchtime and suppertime, each test lasting for 40 minutes.
  Body temperature will be measured during lunch using a thermal imager（Fluke RSE600）in centigrade(℃).

CONTACTS AND LOCATIONS:
Overall Officials: John Speakman, Study Chair — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No